CLINICAL TRIAL: NCT01924416
Title: A Decision Aid With Health-Related Quality of Life (HRQL) Assessment to Reduce Costs in the Treatment of Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Lung Cancer Information Study (LCIS-R01)
Acronym: LCIS-R01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Patricia Hollen, Professor, School of Nursing, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16005; R01CA157409-01A1 (NIH)
Record Dates: First submitted 2013-08-09; First posted 2013-08-16 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Care (Experimental): Enhanced Care: Decision aid; QL-PRO immediate summary results; chemotherapy cycles and imaging studies as needed
  Interventions: Behavioral: Enhanced Care (intervention group and comparison group)
- Usual Care (Active Comparator): Usual Care: Routine chemotherapy cycles and imaging studies
  Interventions: Behavioral: Usual care (routine chemotherapy cycles and imaging studies)

INTERVENTIONS:
Behavioral: Enhanced Care (intervention group and comparison group) — Decision aid coupled with immediate QL-PRO results
  Arms: Enhanced Care
Behavioral: Usual care (routine chemotherapy cycles and imaging studies) — Usual care does not receive intervention
  Arms: Usual Care

SUMMARY:
The primary specific aim is to test the hypothesis that use of a decision aid to enhance informed, shared decision making coupled with quality of life assessment in patients with advanced lung cancer receiving first-, second-, or third-line therapy will lead to a reduction in two major contributors of cost (number of chemotherapy cycles; number of advanced imaging studies) compared with the control arm.

DETAILED DESCRIPTION:
Appropriate utilization of treatment with systemic therapy remains problematic in advanced lung cancer. A major issue continues to be over-treatment. Contributors to this include barriers in communication concerning patients' wishes and goals, lack of formal monitoring of symptoms using validated health-related quality of life (QL) and patient reported outcomes (PROs) assessment, and over-dependence on imaging studies as the major and often sole assessment tool. All of these factors make quality decision making more difficult and can lead to decisional conflict and patient and family regret with treatment. The primary specific aim is to test the hypothesis that use of a decision aid to enhance informed, shared decision making coupled with QL assessment with immediate results in patients with advanced lung cancer receiving first, second, or third-line therapy will lead to a reduction in two major contributors of cost (number of chemotherapy cycles administered and the number of advanced imaging studies [CT, MRI, PET] related to treatment decisions) compared with the control arm. Secondary aims are: 1) To test the hypothesis that patients with advanced lung cancer who receive an intervention decision aid coupled with immediate QL-PRO results) will have reduced decisional conflict, and reduced decisional regret related to the decision-making process, than those who do not; and 2) to explore the hypothesis that patients with advanced lung cancer who have greater agreement with their chosen supporter (less difference in perception of QL-PROs between the patient and the supporter) will have fewer chemotherapy cycles, than those who do not have close agreement. This phase III, two-arm, prospective, randomized clinical trial (RCT) will test the use of a decision aid ("DecisionKEYS") for patients with advanced lung cancer and coupled with the validated, Electronic Lung Cancer Symptom Scale ("eLCSS-QL") to provide immediate QL-PRO results over the treatment period. A repeated measures design will obtain QL assessment at baseline, every 3 weeks while chemotherapy is given, and at the completion of chemotherapy. This study will use a pretest/ posttest design covering timing for each of three consequential decisions of cancer chemotherapy: Decision 1 ("Starting Chemotherapy"), Decision 2 ("Changing Chemotherapy"), and Decision 3 ("Stopping Anti-Cancer Treatment"). There will be three entry points: patients can be entered into the trial either at their initial chemotherapy, or at the time of starting 1st-, 2nd- or 3rd-line chemotherapy. A stratified block randomization design will be used in which strata are determined by two variables: line of therapy and presenting quality of life. This RCT will be conducted in the outpatient setting at three cancer centers in three states. The sample will include 196 patients with advanced non-small cell lung cancer and their chosen supporter (if available). The sampling plan will include serially screening the clinic appointment roster in the clinics. QL-PRO assessment, decisional conflict, and decisional regret will be used to evaluate response to the decision aid. A specific protocol will be followed by the physician and study nurse at each visit. Descriptive statistics, subgroup analyses (t-test), and Generalized Linear Model (GLM) method will be used for analyses.

ELIGIBILITY:
A. Inclusion criteria for lung cancer subject:

1. Pathologically or cytologically determined non-small cell lung cancer (NSCLC)
2. Receiving either first-line, second-line, or third-line chemotherapy for advanced NSCLC. Any chemotherapy will be acceptable
3. Stage IIIB or IV
4. Performance status of KPS 60-100% or ECOG 0-2
5. Hematologic and metabolic parameters suitable for chemotherapy
6. Patients previously treated with adjuvant therapy who now have recurrent NSCLC, will be included as receiving first line therapy
7. Patients with brain metastasis are eligible provided: they are at least 1 week from completion of surgery or RT for brain metastasis, have stable and adequate neurological status to proceed with chemotherapy, and meet all other eligibility criteria
8. Patients with prior cancer diagnoses (with or without prior chemotherapy), are eligible provided the previous malignancy is well controlled
9. Ages greater than 18 with NSCLC
10. Life expectancy greater than three months
11. Able to understand English or Spanish, but is not required to be literate

B. Exclusion criteria for lung cancer subject:

1. Patients treated with molecular targeted therapy as their sole treatment
2. Patients with documented severe psychiatric diagnoses from the medical record, which may prevent full study participation
3. Patients receiving protocol chemotherapy that mandates either the number of cycles of treatment to be received or a fixed schedule of imaging studies
4. Patients receiving concomitant chemotherapy and radiation therapy are not eligible for this protocol
5. Patients who are prisoners
6. Patients who are pregnant (self reporting by patient)
7. Patients who are cognitively impaired

C. Inclusion criteria for supporter:

1. Ages greater than 18
2. Able to understand English or Spanish, but is not required to be literate

D. Exclusion criteria for supporter:

1. Prisoners
2. Patients who are cognitively impaired

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2012-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
A reduction in two major contributors of cost: Number of chemotherapy cycles, and number of advanced imaging studies | 9 weeks
  Number of chemotherapy cycles administered and number of advanced imaging studies (CT, MRI, PET) related to treatment decisions

SECONDARY OUTCOMES:
QL-PRO assessment | Every three weeks for 3 cycles, an expected average of 9 weeks
  Change in QL-PRO assessment at each new cycle to help in informed, shared decision making
Decisional conflict | Pre-post each of three decisions during chemotherapy treament, an expected average of 10 months
  Change in decisional conflict for three treatment decisions:
  Decision 1 (Starting Chemotherapy); Decision 2 (Changing Chemotherapy); Decision 3 (Stopping Anti-Cancer Treatment)
Decisional regret | Post each of three decisions during chemotherapy treatment, an expected average of 10 months
  Degree of decisional regret after each of three treatment decisions:
  Decision 1 (Starting Chemotherapy); Decision 2 (Changing Chemotherapy); Decision 3 (Stopping Anti-Cancer Treatment)
Overall decisional regret | 1-2 weeks followup at end of chemotherapy treatment, an expected average of 10 months
  Degree of decisional regret after completion of treatment (1-2 weeks followup telephone contact)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J Hollen, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States